CLINICAL TRIAL: NCT03891069
Title: Feasibility and Safety of the AHA Exergame System in Parkinson's Disease Patients: a Mixed Methods Study
Brief Title: Feasibility of the AHA Exergame System in Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Neurológico Sénior (Other)
Collaborators: University of Lisbon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CNS2019-01
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Exergames; Virtual reality; Exercise; Feasibility study
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: A mix-methods study, including two focus groups (with patients and physiotherapists) and quantitative feasibility study, will performed. Physiotherapists and PD patients with a Hoehn Yahr Stage ≤ 2 (MED ON), ability to walk independently without risk of falling and a Mini-mental state score > 24 will be included. The primary outcome will be patients' satisfaction with the games measured through a 7-point Likert scale. Secondary outcomes will include: games difficulty (7-point Likert scale), perceived effort (modified Borg scale), safety (number of adverse events) and functional mobility (Time up and Go test).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Participants will be invited to play the five different Exergames, for a total of 5 minutes.
  Interventions: Device: AHA Exergame System

INTERVENTIONS:
Device: AHA Exergame System — The AHA Exergame System consists of a mobile computing platform running a set of parameterizable exergames purposely designed for elderly fitness training. The platform is equipped with a 1000 lumens video projector capable of creating a 2.05m by 1.16m floor projection display and a Kinect V2 sensor to serve as game controller. The AHA exercise-based computer games have been designed for and tested with elderly people and were adapted for the functional limitations of PD patients. The system includes five different games that aim to train patients motor ability, cardiorespiratory and muscular strength.

SUMMARY:
Background: Parkinson's disease (PD) remains a progressive disease associated with a high level of disability. Due to the physical and cognitive impairments, fatigue and apathy, patients frequently experience a decrease in their daily physical activity. Exercise programs have been recommended for symptomatic control, however, its implementation is still challenging in terms of acceptability and adherence. Exergames (i.e. exercise based on video games) have been proposed as a potential, home-based rehabilitation tool to improve PD patients motor skills and to promote a more active lifestyle.

Methods: This study aims to evaluate the feasibility and safety of an exergames system design for PD patients' rehabilitation. A mix-methods study, including two focus groups (with patients and physiotherapists) and quantitative feasibility study, will be performed. Physiotherapists and PD patients with a Hoehn Yahr Stage ≤ 2 (MED ON), ability to walk independently without risk of falling and a Mini-mental state score > 24 will be included. The primary outcome will be patients' satisfaction with the games measured through a 7-point Likert scale. Secondary outcomes will include games difficulty (7-point Likert scale), perceived effort (modified Borg scale), safety (number of adverse events) and functional mobility (Time up and Go test).

DETAILED DESCRIPTION:
1. Background Parkinson's disease (PD) is a neurological disorder, characterized by the presence of motor and non-motor symptoms that negatively affects patients' quality of life. (1,2) Despite optimal medical treatment, patients develop a progressive disability that usually shapes a sedentary lifestyle, which is a risk factor for cardiovascular disease, diabetes mellitus, cognitive impairment, osteoporosis, and depression. (1,3,4) In the past years, physiotherapy and exercise have been recommended for symptomatic control and as a strategy to reverse PD patients' sedentary lifestyles. (2,5) However, results from previous studies showed that physiotherapy programs only provide a short-term benefit and it still a challenge the implementation of unsupervised home-based exercise. (3,6) Exergames are video games to exercise, based on gross physical movements of the player, that combine real-time motion detection with engaging games. (7,8) They have been described as a therapeutic tool that includes functional, purposeful and appealing exercise, with positive effects in neurological diseases and older adults. (7,8) Exergames promote an integrated motor and cognitive stimulation, providing biofeedback, enhancing game performance and learning of the virtual tasks with transference to real conditions and its home-based characteristics. Based on this, exergames have been proposed as a complement to physiotherapy programs, in order to improve PD motor symptoms. (7,8) However, they should be specifically tailored to address PD functional needs, in order to optimize efficacy, adherence, and safety. (8) This study aims to evaluate the feasibility and safety of an exergames system design for PD patients.
2. Participants and methods

   Study design A feasibility study including two phases, one qualitative and another quantitative will be performed.

   In the first phase, the qualitative study, two focus groups will be conducted (one with PD patients and other with a group of physiotherapists), to discuss the accessibility and usability of the exergames to be tested and the exercise-based computer games for people with PD. The second phase, the quantitative study, will be a single-center, open-label, feasibility, and usability study.

   Patients recruitment PD patients will be recruited from the Campus Neurológico Sénior (CNS) institution to participate either in the qualitative phase or in the quantitative phase. Patients will be included if they were: 1) idiopathic PD patients according to the UKBB criteria; 2) age between 40-80 years old; 3) with a Hoehn Yahr Stage (HY) 1 or 2 in MED ON; 4) ability to walk independently without risk of falling; 5) a Mini-mental state score > 24; 6) ability to communicate with the investigator, to understand and comply with the requirements of the study; and lastly 7) ability to provide written informed consent to participate in the study.

   Patients will be excluded if they had an atypical parkinsonian syndrome. Physiotherapists will be also screened and recruited from the CNS institution. The Local Ethical Committee approved the study (Ref. 9/2017). All included patients and physiotherapists will provide informed consent, before enrolling in any study procedure.

   Intervention and assessment The AHA Exergame System consists of a mobile computing platform running a set of parameterizable exergames purposely designed for elderly fitness training. The platform is equipped with a 1000 lumens video projector capable of creating a 2.05m by 1.16m floor projection display and a Kinect V2 sensor to serve as game controller.(9) The AHA exercise-based computer games have been designed for and tested with elderly people and were adapted for the functional limitations of PD patients. The system includes five different games that aim to train patients motor ability, cardiorespiratory and muscular strength.

   Patients Focus groups The focus group will be conducted using a semi-structured script where participants will be asked to discuss their thoughts on Exergames, daily use of technology and preferences for the style and type of games.

   During the session, participants will be invited to view and play with the five games to have their perception of the appropriateness of the games for people with PD. This part of the focus group will be followed by a member of the IT team and a physiotherapist to provide support for instructions guidance and to guarantee the participant's safety while trying the games. In the end, patients will be asked to share their thoughts on which features they would like to see included in the proposed games.

   The focus group will be recorded, with the agreement of all participants, to be transcribed for inductive thematic qualitative analysis.

   Physiotherapists focus groups The focus group will be developed using a semi-structured script where the physiotherapists' participants will be asked for their opinion on Exergames, the usability of this tool during the sessions, advantages, and disadvantages.

   During the focus group, physiotherapists will be invited to play the games to comment on the features presented and its adequacy to PD patients. At this point, a member of the IT team will provide support at a technical level and for instructions guidance.

   The focus group will be recorded, with the agreement of all participants, to be transcribed for inductive thematic qualitative analysis.

   Quantitative study Baseline assessment Before any data will be recorded, each patient reviewed and signed an informed consent form. In order characterize the sample, demographic data (date of birth, age, gender, height, weight) and medical history (age of onset, disease duration, medication) will be collected, and three rating scales and clinical tests (MDS-UPDRS, HY and Time Up and Go (TUG) test) administered.

   Intervention Participants will be invited to play the five different Exergames. Before playing the games, each participant will have a training period, in which the game will be presented, and the instructions explained. The sequence in which the games will be played will be randomized using computer software. Each game will be played for a total time of 5 minutes. In the end, patients will rate their satisfaction with the game and its difficulty through a 7-point Likert scale and the perceived exertion through a modified Borg scale. At the end of the intervention, the TUG test followed by the modified Borg scale will be repeated.

   Exergames overview

   Grape Stomping (Douro Region) - Cardiorespiratory Training The goal of this Exergame is to stomp on grapes, pulled from the conveyor belt into the tank by dragging small virtual grape baskets. To do that, flexion-extension arm movements are needed to drag the grape bunches into the tanks, once done, the stomping process starts, requiring users to raise the knees to a pre-defined height to produce the wine. After fill up one of the tanks, users are asked to move to the others to continue the exercise. The experience ends once the pre-established training time finalizes, thus screening the number of tanks filled, the number of litres of wine produced, the number of steps performed and the number of grape bunches dragged.

   Rabelos VR (Porto City) - Upper limbs, Muscular Strength Training The goal of this Exergame is to row along the river collecting several wine barrels located in small docks at the river banks. Users are encouraged to make circular arm movements simulating rowing gestures to move the boat forward. For the lateral displacements of the boat, users can be standing and use lateral movements or trunk leaning; or they can be seated using trunk leaning. Additionally, to navigate the treacherous rapids, users have to avoid big rocks randomly located in the riverbed while trying to dock on the margins to pick up one or multiple wine barrels. To do that, users must turn the trunk to the side of the dock and make an extension-flexion movement of the elbow to simulate picking up the barrels. Meanwhile, the boat is stopped until users picked up, one by one, all of the barrels in the docks and subsequently the users should The Exergame ends with the countdown of the pre-established time, screening the number of rocks hit, completed rows and collected barrels as well as the time spent rowing and collecting.

   Toboggan Ride (Madeira Island) - Balance, Trunk Muscular Strength The main goal in this Exergame is to successfully collect as much objects as possible in a pre-established time avoiding crashes with cars and pedestrians. The sledge direction is controlled via trunk lateral flexions to the right and to the left while the acceleration is controlled through trunk flexion-extension movements. Flexion movements are used to increase the acceleration of the vehicle while extensions are used to deaccelerate it. Collecting and crashing events occur when the virtual vehicle make a collision with each individual object making specific rewarding/punishment game sounds. The journey finalizes with a screenshot of metrics encompassing the time of the session and the number of objects collected.

   Exerfado (Lisbon City) - Lower Limbs, Muscular Strength Training The main objective is the user to collect each musical note by positioning him/herself in front of the note trajectory. Additionally, the user needs to "push" wrong notes that are sliding in the wrong trajectory and then collect them equally at the right position. Collecting the right notes at the right position will reward the user by incrementing the percentage of notes collected. Some notes are special and offer extra bonus, they are identified in the game with a glowing and sparking effect. The wrong notes are displayed in game with black color and with a blinking arrow indicating the direction to where needs to be pushed, if the user is able to perform the correct arm gesture before the musical note is lost, the wrong note changes to the correct trajectory and to the right color. Notes are pushed with arm extension which can be predefined as low or high. User has to move left and right within the projection range. A piano key is represented as "pressed" when the user is in front of it and indicates that a note coming in that trajectory will be collected. User position can be tracked by the waist joint or by both feet; in this case the user will be able to select two piano keys at the same time. Interaction ends when the music stops playing.

   To better adapt to each user needs, on the configuration menu is possible to change settings such as arm extension, joint to be tracked, the percentage of notes, note sliding time, and musical choice from a list.
3. Statistical methods and data analysis

   Sample size

   Qualitative Study For the focus group, 5 PD patients will be invited to participate in the qualitative study. For the physiotherapist approach, 5 participants will be invited with experience in dealing with PD patients.

   Quantitative Study Assuming this is an exploratory study, there is no rationale to estimate the sample size, a total of 10 participants will be asked to participate in the quantitative phase, with the condition they did not take part of the qualitative phase.

   Data Analysis A content analysis will be performed on the qualitative data assuming a deductive approach. The content analysis will be performed using a descriptive and interpretative analysis of the focus group.

   The statistical analysis for the qualitative phase of the study will be performed using SPSS® version 21.0; SPSS Inc. Chicago, IL. Data will be described using descriptive statistics.

   As our primary outcome, we will measure patients' satisfaction with the games, through a 7-point Likert scale, at the end of each game and at the end of the intervention (global perspective).

   The secondary outcomes will be:
   * Patients level of difficulty with the game measures through a 7-point Likert scale;
   * Changes in the level of perceived exertion measure at the end of each game and from baseline to end of all games with the modified Borg scale;
   * Number of adverse events;
   * Changes in the TUG test result from baseline to end of the intervention.
4. Safety issues and adverse events reporting Adverse events will be collected for the duration of the study and at the Follow-Up visit. It is not expected that participation in the study will be associated with risks or will increase the risk of adverse effects. All therapeutic interventions will be recommended to be kept stable.

   Research subjects will be questioned about adverse events during the Clinical Assessment and follow up visit. All adverse events (serious or non-serious) and any other abnormal clinical findings will be recorded in the subjects' case report form (CRF). For all adverse events, sufficient information will be pursued to permit:
   * a determination of a temporal relationship;
   * an adequate determination of the outcome of the event (i.e., whether the event should be classified as a serious adverse event);
   * an assessment of the causal relationship between the adverse event and the study requirements.

   An abnormal result finding will be classified as an adverse event if one or more of the following criteria are met:
   * The resulting finding leads to discontinuation of subject participation in the research study;
   * The resulting finding is considered an adverse event by the researcher.
5. Withdrawal of subjects Subjects will be able to withdrawal from the study at any time of the research study. After withdrawal, no more data will be collected and taken into consideration for statistical purposes regarding the withdrawal subjects.

Withdrawal criteria will include, for example: adverse events (serious and non-serious), lack of compliance to testing, subject fails to comply with protocol requirements, subject's voluntary withdrawal of consent.

Replacements will not be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson's disease according to MDS criteria
* Age ≥ 40 and ≤ 80 years old
* Hoehn and Yahr stages between I, II and III (MED ON)
* MMSE > 24
* Ability to walk independently without risk of falling
* Ability to communicate with the investigator, to understand and comply with the requirements of the study
* Willing and able to provide written informed consent to participate in the study
* Being interested in participating in this study

Exclusion Criteria:

* Patients diagnosed with atypical parkinsonian syndromes
* Significant postural instability in ON likely to affect gait and/or have the need to use a walking aid to walk safely
* Presence of severe dyskinesia's
* Having any other neurological/orthopedic disorders likely to affect gait, e.g., history of stroke
* Having significant active psychiatric problems (example: hallucinations, confusion, psychosis) that aggravates patient´s symptoms when dealing with the use of -Exergames
* Inability to correctly respond to the assessment protocol according to the clinician's judgment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Patients' satisfaction with the games | End of each game and at the end of the intervention, up to 5 hours after baseline assessment
  Patients' satisfaction with the games, through a 7-point Likert scale, at the end of each game and at the end of the intervention (global perspective)

SECONDARY OUTCOMES:
Level of difficulty | End of each game and at the end of the intervention, up to 5 hours after baseline assessment
  Patients level of difficulty with the game measures through a 7-point Likert scale
Level of perceived exertion | End of each game and at the end of the intervention, up to 5 hours after baseline assessment
  Changes in the level of perceived exertion measure at the end of each game and from baseline to end of all games with the modified Borg scale
Number of adverse events | Up to 2 days after baseline assessment
  Frequency of adverse events during study period
Efficacy on functional mobility | Baseline and end of the intervention, up to 5 hours after baseline assessment
  Changes in TUG test result from baseline to end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Ferreira, MD, PhD, Principal Investigator — Campus Neurológico Sénior
Locations (1):
- Campus Neurológico Sénior, Torres Vedras, Portugal